CLINICAL TRIAL: NCT04716608
Title: Treatment for Osgood Schlatter Patients With a Physiotherapy Program "TrOPhy-Study"
Brief Title: Treatment for Osgood Schlatter Patients With a Physiotherapy Program
Acronym: TrOPhy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-02132; ks20Neuhaus
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Osgood-Schlatter Disease
Keywords: myofascial massage; stretching; home exercises; strengthening; KOOS-Child-Questionnaire
MeSH Terms: conditions — Osteochondrosis

STUDY DESIGN:
Intervention Model Description: randomised controlled parallel groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 INT (= intervention) (Active Comparator): physiotherapy program with
  * Myofascial Release Massage (quadriceps)
  * Foam Rolling lower extremity
  * Knee Isometrics in knee extension (sitting position)
  * Dynamic and static stretching (quadriceps) in half knee position
  * Core Stability (planks)
  * Strengthening (calf raises, good morning,squats, squat jump)
  * Balance (single leg stance)
  Interventions: Other: physiotherapy program
- Group 2 USC (= usual care) (Placebo Comparator): usual care treatment with
  * Core Stability (prone plank)
  * Strengthening: (Hip extension, abduction; Calf raises)
  * Stretching (M. rectus femoris (static) in standing position; Hamstring in sitting position)
  * Balance (single leg stand)
  Interventions: Other: usual care treatment

INTERVENTIONS:
Other: physiotherapy program — physiotherapy program with Myofascial Release Massage, stretching, strengthening.
  2 sessions per week (duration 30 minutes per session) for 8 weeks, supervised by a physiotherapist; complemented by a home training program.
  Arms: Group 1 INT (= intervention)
Other: usual care treatment — stretching,strengthening; 2 sessions per week (duration 30 minutes per session) for 8 weeks
  Arms: Group 2 USC (= usual care)

SUMMARY:
This study is to compare the effect of a physiotherapy program to usual care treatment in patients with Osgood Schlatter disease (OSD). Patients will be randomly assigned into two groups. Group 1 will receive the physiotherapy program with myofascial massage, while group 2 (usual care group USC) will receive usual care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral OSD
* ability to follow instructions
* sufficient knowledge of German
* availability: can participate in two exercise sessions per week for a period of 8 weeks

Exclusion Criteria:

* any history of knee surgery
* medication intake affecting the knee
* unstable fractures
* neurological disorders
* systematic diseases
* already in physiotherapeutic treatment because of the knee
* not possible to do any physiotherapy sessions at the Universitäts-Kinderspital Basel (UKBB)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
change in Knee and Osteoarthritis Outcome Score for Children (KOOS-Child-Questionnaire Score) | at baseline and 8 weeks after baseline
  KOOS-Child is a patient-reported outcome measure employing five-item Likert scales. KOOS-Child covers 5 dimensions (subscales): Pain, Symptoms (titled "Knee problems" in the KOOS-Child), Difficulty during daily activities (ADL), Function in sport and play (Sports/Play) and knee-related Quality of Life (QOL). 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems

SECONDARY OUTCOMES:
Change in Knee pain assessed by Visual Analogue Scale (VAS) | at baseline and 8 weeks after baseline
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, 10 cm in length, with the left side signifying no pain and the right side signifying the worst pain ever.
Change in Range of motion (ROM) of knee | at baseline and 8 weeks after baseline
  Range of motion is typically measured using a goniometer. Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Y Balance Test (Lower Quarter) | at baseline and 8 weeks after baseline
  The Y-Balance Test is a dynamic test performed in a single-leg stance that requires strength, flexibility, core control and proprioception. The goal of this test is to maintain single-leg balance on one leg while reaching as far as possible with the contralateral leg in three different directions. The three movement directions are anterior, posteromedial and posterolateral, performed on each leg. Each test is repeated three times, and the maximum reach in each direction is recorded.
Time of return to sport activity (in days) | within 8 weeks after baseline
  Time of return to sport activity (in days) since start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Faude, PD Dr. med., Principal Investigator — Department of Sport, Exercise and Health, Medical Faculty University of Basel
Locations (1):
- Department of Sport, Exercise and Health, Medical Faculty University of Basel, Basel, Switzerland